CLINICAL TRIAL: NCT06835309
Title: Implications of Isokinetic Strengthening of Hip Muscles on Pelvic Floor Muscles Function in Women Experiencing Stress Urinary Incontinence
Brief Title: Isokinetic Strengthening of Hip Muscles Effect on Pelvic Floor Muscles Function in Females With SUI
Acronym: SUI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005601
Record Dates: First submitted 2025-01-23; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Isokinetic Strengthening; Pelvic Floor Muscles; Stress Urinary Incontinence (SUI)
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Pelvic floor muscles exercises
  Interventions: Other: Pelvic floor muscles exercises
- Treatment arm (Experimental): Pelvic floor muscles exercises and isokinetic strengthening of hip muscles
  Interventions: Other: Pelvic floor muscles exercises and isokinetic strengthening of hip muscles

INTERVENTIONS:
Other: Pelvic floor muscles exercises — The exercises for strengthening the PFM were 10 contractions of 5 seconds, 15 contractions of 3 seconds, 20 contractions of 2 seconds, 20 contractions of 1 second (equal rest time between contractions), and 5 repetitions of maximum contractions while coughing (1-minute interval).25 The level of difficulty of the exercises throughout the 20 sessions was determined by the patient's position, starting in a supine position, then progressing to a sitting position and, finally, to a standing position
  Arms: Control arm
Other: Pelvic floor muscles exercises and isokinetic strengthening of hip muscles — The hip muscle strengthening exercise was executed on Biodex multi-joint system isokinetic dynamometer. Muscle tension of the lower limbs was relieved by executing 5-minute warm-up exercises using a cycle ergometer before execution of the isokinetic exercise For each hip muscle group, eight repetitions per set for 4 sets were carried out for a single exercise with a 30 second break between each set. The patient's position were the same positions used in the testing procedure. The exercises were carried out 3 times a week and the hip muscles strength evaluation was conducted after the end of the program intervention
  Arms: Treatment arm

SUMMARY:
This study will be conducted to investigate the impact of isokinetic strengthening of hip muscles on pelvic floor muscles function in women experiencing stress urinary incontinence Does isokinetic strengthening of hip muscles impact pelvic floor muscles function in women experiencing stress urinary incontinence?

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stress urinary incontinence
* age between 30 and 50 years

Exclusion Criteria:

* low back pain
* lower limb muscle pathology and/or joint degeneration
* cardiovascular, metabolic or pulmonary disease
* body mass index (BMI) > 30 kg/m2.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-04-23 (Estimated); Study Completion 2025-05-23 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle strength | 12 weeks
  Perineometry to measure vaginal squeeze pressure (in mm hg) the more the grade, the better the muscle strength and so the less the stress urinary incontinence

SECONDARY OUTCOMES:
Stress urinary incontinence. | 12 weeks
  - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) to evaluate the frequency, severity and impact on quality of life) the less the grade, the better the muscle strength and so the less the stress urinary incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/